CLINICAL TRIAL: NCT05218733
Title: Postoperative Analgesia in Patients Undergoing Total Abdominal Hysterectomy: A Randomized Controlled Comparison Between Ultrasound Guided Erector Spinae Plane Block and Intrathecal Morphine
Brief Title: Ultrasound Guided Erector Spinae Plane Block vs Intrathecal Morphine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ibrahim Mamdouh Esmat, Assistant Professor of Anesthesia and Intensive Care Department, Faculty of Medicine, Ain-shams University, Cairo, Egypt., Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB 00006379//31-1-2022
Record Dates: First submitted 2022-01-31; First posted 2022-02-01 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- G1 Group: (Erector Spinae Plane Block (ESPB) Group) (Active Comparator)
  Interventions: Procedure: Ultrasound Guided Erector Spinae Plane Block
- G2 Group: (Intra thecal morphine (ITM) Group) (Active Comparator)
  Interventions: Drug: Intra thecal morphine.
- G3 Group: (Control Group) (Other)
  Interventions: Drug: General anesthesia using intravenous fentanyl (1µgm/kg)

INTERVENTIONS:
Procedure: Ultrasound Guided Erector Spinae Plane Block — General anesthesia using intravenous fentanyl (1µgm/kg) and patients will receive bilateral ultrasound-guided ESPB by the an experienced anesthetist in US regional blocks, with each block 20 mL of bupivacaine 0.25%
  Arms: G1 Group: (Erector Spinae Plane Block (ESPB) Group)
Drug: Intra thecal morphine. — General anesthesia using intravenous fentanyl (1µgm/kg) and patients will receive intra thecal morphine with spinal needle 25G, 3 ml containing 300 ug preservative free morphine
  Arms: G2 Group: (Intra thecal morphine (ITM) Group)
Drug: General anesthesia using intravenous fentanyl (1µgm/kg) — Patients will receive general anesthesia using intravenous fentanyl (1µgm/kg)
  Arms: G3 Group: (Control Group)

SUMMARY:
Total abdominal hysterectomy (TAH) is a major surgical procedure after which significant post-operative pain and discomfort are anticipated. Abdominal field blocks have been followed for many years and extensively used for pain management following abdominal surgeries such as laparotomies and appendicectomies. Erector Spinae Plane Block (ESPB)-first recently described for the treatment of thoracic neuropathic pain, is a peri-paravertebral regional anesthesia technique that has since been reported as an effective technique for prevention of postoperative pain in various surgeries. Intrathecal opioid administration is an attractive analgesic technique since the opioid is injected directly into the cerebrospinal fluid, close to the structures of the central nervous system where the opioid acts.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) 25 to 35kg/m².
* American Society of Anesthesiologist (ASA) physical status I or II.

Exclusion Criteria:

* patient's refusal
* Altered mental status
* Known allergy to study drugs (bupivacaine or morphine)
* Local infection at site of puncture.
* Known case with any pulmonary disease
* Known case with Obstructive sleep apnea (OSA)
* Coagulopathy and /or thrombocytopenia
* Chronic pain
* Severe hepatic or kidney impairment

Ages: 40 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
The time for requirement of first rescue analgesic (min) | 24 hours postoperatively
  The time for requirement of first rescue analgesic (min)

CONTACTS AND LOCATIONS:
Locations (1):
- Ain-Shams University Hospitals, Cairo, Egypt

REFERENCES:
- [Derived] Ashoor TM, Esmat IM, Algendy MA, Mohamed NR, Talaat SM, Rabie AH, Elsayed AM. Comparison of the postoperative analgesic efficacy of the ultrasound-guided erector spinae plane block and intrathecal morphine in patients undergoing total abdominal hysterectomy under general anesthesia: a randomized controlled trial. J Anesth. 2025 Apr;39(2):299-310. doi: 10.1007/s00540-025-03466-1. Epub 2025 Mar 6. PMID 40047853